CLINICAL TRIAL: NCT05336500
Title: Effectiveness of Education to Keep the Abdomen Relaxed Versus Contracted During Pilates Exercises in Patients With Primary Chronic Low Back Pain: a Randomised Controlled Trial
Brief Title: Effectiveness of Education to Keep the Abdomen Relaxed Versus Contracted During Pilates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitário Augusto Motta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KAR/KAC
Record Dates: First submitted 2022-04-12; First posted 2022-04-20 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2022-10

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates method exercises associated with education to keep the abdomen relaxed (Experimental): The group will receive guidance to perform the exercises in a relaxed and smooth way
  Interventions: Other: Pilates method exercises
- Pilates method exercises associated with education to keep the abdomen contracted (Active Comparator): The group will receive guidance on the specific activation of the center of strength (the powerhouse)
  Interventions: Other: Pilates method exercises

INTERVENTIONS:
Other: Pilates method exercises — Participants will be randomised into two groups that will be treated with Pilates exercises for 12 weeks (twice a week for 60 minutes). The control group will receive guidance on the specific activation of the center of strength (the powerhouse), while the experimental group will receive guidance to perform the exercises in a relaxed and smooth way.

SUMMARY:
This study aims to investigate the effectiveness of education to keep the abdomen relaxed versus contracted during Pilates exercises in patients with primary chronic low back pain.

Participants will be randomised into two groups that will be treated with Pilates exercises for 12 weeks. The control group will receive guidance on the specific activation of the center of strength (the powerhouse), while the experimental group will receive guidance to perform the exercises in a relaxed and smooth way. Primary outcomes will be pain intensity and disability 12 weeks post randomisation.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 years old;
* Low back pain for more than 3 months;
* Disability level ≥ 4 points on the Roland-Morris Disability Questionnaire (RMDQ);
* Ability to move independently with or without assistance;
* Ability to understand Portuguese enough to be able to fill in the questionnaires.

Exclusion Criteria:

* The main area of pain other than the lumbar spine (eg, nerve root compression or herniated disc with radicular pain, lateral or central stenosis);
* Surgery performed on the lumbar spine.
* Surgery performed on the lower limbs, or abdominal region less than 6 months ago;
* Performing an invasive procedure for pain relief (eg, epidural injection, rhizotomy) in the last 3 months;
* Diagnosis of inflammatory rheumatologic diseases, progressive neurological disease, or viral diseases as the primary cause of pain;
* Scoliosis as the primary cause of pain;
* Unstable heart conditions;
* Presence of red flags such as malignancy/cancer, acute trauma (less than 6 months), infection, spinal cord/cauda equina compression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 12 weeks post randomisation
  Pain intensity will be obtained through self-report by the Brazilian version of the 11-point Numerical Pain Scale (NPS) (Costa et al., 2008; Vigotsky et al., 2021), which varies between 0 and 10 points, where 0 is "no pain" and 10 is "the worst pain imaginable" where individuals should report pain intensity based on the last 7 days.
Disability related | 12 weeks post randomisation
  Disability will be obtained through self-report by the Brazilian version of the Roland-Morris Disability Questionnaire (RMDQ) (Nusbaum et al., 2001), which has 24 statements involving activities and pain situations, to which the patient is instructed to answer "yes" only to those described in the assessment day, and each answer corresponds to one point.

SECONDARY OUTCOMES:
Perception of global improvement | 12 weeks post randomisation
  Perception of global improvement will be obtained through self-report by the Perception of Global Effect Scale (PGES), 11 points ranging from -5 ("much worse"), 0 ("no change") to +5 (completely recovered) (Costa et al., 2008). For all measures of perceived global effect participants will be asked: "Compared to the start of your first episode, how do you describe your low back pain in the past few days?". A highly positive score indicates greater recovery, while a negative score indicates worsening of symptoms.
Specific functionality | 12 weeks post randomisation
  Specific functionality will be obtained through self-report by the Patient-specific functional scale (PSFS) (Costa et al., 2008), which consists of an interview in which the patient chooses three important activities whose execution is difficult or impossible due to low back pain. For each activity, a score of difficulty ranges from 0 (unable to perform) to 10 (able to perform at the same level as before the problem).

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Universitário Augusto Motta, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Costa LO, Maher CG, Latimer J, Ferreira PH, Ferreira ML, Pozzi GC, Freitas LM. Clinimetric testing of three self-report outcome measures for low back pain patients in Brazil: which one is the best? Spine (Phila Pa 1976). 2008 Oct 15;33(22):2459-63. doi: 10.1097/BRS.0b013e3181849dbe. PMID 18923324
- [Background] Nusbaum L, Natour J, Ferraz MB, Goldenberg J. Translation, adaptation and validation of the Roland-Morris questionnaire--Brazil Roland-Morris. Braz J Med Biol Res. 2001 Feb;34(2):203-10. doi: 10.1590/s0100-879x2001000200007. PMID 11175495
- [Background] Vigotsky AD, Tiwari SR, Griffith JW, Apkarian AV. What Is the Numerical Nature of Pain Relief? Front Pain Res (Lausanne). 2021 Nov 2;2:756680. doi: 10.3389/fpain.2021.756680. eCollection 2021. PMID 35295426
- [Background] Campbell A, Kemp-Smith K, O'Sullivan P, Straker L. Abdominal Bracing Increases Ground Reaction Forces and Reduces Knee and Hip Flexion During Landing. J Orthop Sports Phys Ther. 2016 Apr;46(4):286-92. doi: 10.2519/jospt.2016.5774. Epub 2016 Mar 8. PMID 26954271
- [Background] Coenen P, Campbell A, Kemp-Smith K, O'Sullivan P, Straker L. Abdominal bracing during lifting alters trunk muscle activity and body kinematics. Appl Ergon. 2017 Sep;63:91-98. doi: 10.1016/j.apergo.2017.04.009. Epub 2017 Apr 22. PMID 28502411
- [Background] Eliks M, Zgorzalewicz-Stachowiak M, Zenczak-Praga K. Application of Pilates-based exercises in the treatment of chronic non-specific low back pain: state of the art. Postgrad Med J. 2019 Jan;95(1119):41-45. doi: 10.1136/postgradmedj-2018-135920. Epub 2019 Jan 12. PMID 30636192
- [Background] Foster NE, Anema JR, Cherkin D, Chou R, Cohen SP, Gross DP, Ferreira PH, Fritz JM, Koes BW, Peul W, Turner JA, Maher CG; Lancet Low Back Pain Series Working Group. Prevention and treatment of low back pain: evidence, challenges, and promising directions. Lancet. 2018 Jun 9;391(10137):2368-2383. doi: 10.1016/S0140-6736(18)30489-6. Epub 2018 Mar 21. PMID 29573872
- [Background] Fuhro FF, Fagundes FRC, Manzoni ACT, Costa LOP, Cabral CMN. Orebro Musculoskeletal Pain Screening Questionnaire Short-Form and STarT Back Screening Tool: Correlation and Agreement Analysis. Spine (Phila Pa 1976). 2016 Aug 1;41(15):E931-E936. doi: 10.1097/BRS.0000000000001415. PMID 26720177
- [Background] Gubler D, Mannion AF, Schenk P, Gorelick M, Helbling D, Gerber H, Toma V, Sprott H. Ultrasound tissue Doppler imaging reveals no delay in abdominal muscle feed-forward activity during rapid arm movements in patients with chronic low back pain. Spine (Phila Pa 1976). 2010 Jul 15;35(16):1506-13. doi: 10.1097/BRS.0b013e3181c3ed41. PMID 20431436
- [Background] Hartvigsen J, Hancock MJ, Kongsted A, Louw Q, Ferreira ML, Genevay S, Hoy D, Karppinen J, Pransky G, Sieper J, Smeets RJ, Underwood M; Lancet Low Back Pain Series Working Group. What low back pain is and why we need to pay attention. Lancet. 2018 Jun 9;391(10137):2356-2367. doi: 10.1016/S0140-6736(18)30480-X. Epub 2018 Mar 21. PMID 29573870
- [Background] Hayden JA, Ellis J, Ogilvie R, Malmivaara A, van Tulder MW. Exercise therapy for chronic low back pain. Cochrane Database Syst Rev. 2021 Sep 28;9(9):CD009790. doi: 10.1002/14651858.CD009790.pub2. PMID 34580864
- [Background] Hoffman J, Gabel CP. The origins of Western mind-body exercise methods. Phys Ther Rev. 2015 Nov 2;20(5-6):315-324. doi: 10.1080/10833196.2015.1125587. Epub 2016 Apr 8. PMID 27695277
- [Background] Latey P. The Pilates method: history and philosophy. Journal of Bodywork and Movement Therapies. , 2001; 5: 275-282.
- [Background] Lima M, Ferreira AS, Reis FJJ, Paes V, Meziat-Filho N. Chronic low back pain and back muscle activity during functional tasks. Gait Posture. 2018 Mar;61:250-256. doi: 10.1016/j.gaitpost.2018.01.021. Epub 2018 Mar 20. PMID 29413793
- [Background] Maced, CSG, Debiagi PC, Andrade FM. The Isostretching effect in the muscle strength of gluteus maximus, abdominal and the trunk extensor, incapacity and pain in patients with low back pain. Fisioter. Mov. 2010; 23: 113-120.
- [Background] Maher C, Underwood M, Buchbinder R. Non-specific low back pain. Lancet. 2017 Feb 18;389(10070):736-747. doi: 10.1016/S0140-6736(16)30970-9. Epub 2016 Oct 11. PMID 27745712
- [Background] Mostagi FQ, Dias JM, Pereira LM, Obara K, Mazuquin BF, Silva MF, Silva MA, de Campos RR, Barreto MS, Nogueira JF, Lima TB, Carregaro RL, Cardoso JR. Pilates versus general exercise effectiveness on pain and functionality in non-specific chronic low back pain subjects. J Bodyw Mov Ther. 2015 Oct;19(4):636-45. doi: 10.1016/j.jbmt.2014.11.009. Epub 2014 Nov 18. PMID 26592221
- [Background] Muscolino JE, Cipriani S. Pilates and the "powerhouse." Journal of Bodywork and Movement Therapies. 2016; 8: 15-24.
- [Background] Silva PHB, Silva DF, Oliveira JKS, Oliveira FB. The effect of the Pilates method on the treatment of chronic low back pain: a clinical, randomized, controlled study. Brazilian Journal Of Pain. 2018; 1: 21-28.
- [Background] Sterne JA, White IR, Carlin JB, Spratt M, Royston P, Kenward MG, Wood AM, Carpenter JR. Multiple imputation for missing data in epidemiological and clinical research: potential and pitfalls. BMJ. 2009 Jun 29;338:b2393. doi: 10.1136/bmj.b2393. PMID 19564179
- [Background] Wajswelner H, Metcalf B, Bennell K. Clinical pilates versus general exercise for chronic low back pain: randomized trial. Med Sci Sports Exerc. 2012 Jul;44(7):1197-205. doi: 10.1249/MSS.0b013e318248f665. PMID 22246216
- [Background] Wells C, Kolt GS, Bialocerkowski A. Defining Pilates exercise: a systematic review. Complement Ther Med. 2012 Aug;20(4):253-62. doi: 10.1016/j.ctim.2012.02.005. Epub 2012 Mar 13. PMID 22579438
- [Derived] Lunkes LC, Dias Neto MA, Barra LF, de Castro LR, Ferreira AS, Meziat-Filho N. Education to keep the abdomen relaxed versus contracted during pilates in patients with chronic low back pain: study protocol for a randomised controlled trial. BMC Musculoskelet Disord. 2023 Jan 20;24(1):49. doi: 10.1186/s12891-023-06160-z. PMID 36670384